CLINICAL TRIAL: NCT07104578
Title: Evaluation of the Impact of Pleuropulmonary Ultrasound Performed by the Emergency Physician on the Diagnosis of Dyspnea in the Prehospital Setting
Brief Title: Evaluation of the Impact of Pleuropulmonary Ultrasound on the Diagnosis of Dyspnea
Acronym: LU-SMUR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0219; ID-RCB (Other: 2025-A00990-49)
Record Dates: First submitted 2025-07-07; First posted 2025-08-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Dyspnea
Keywords: dyspnea; pleuropulmonary ultrasound; diagnostic
MeSH Terms: conditions — Dyspnea; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with respiratory distress: patients in respiratory distress treated by the SMUR
  Interventions: Diagnostic Test: Pleuropulmonary ultra sound

INTERVENTIONS:
Diagnostic Test: Pleuropulmonary ultra sound — pleuropulmonary ultrasound performed as part of the treatment

SUMMARY:
Dyspnea is a subjective symptom perceived by the patient as a sensation of "breathing discomfort", "suffocation", "lack of air" or "difficulty inhaling or exhaling". It is a frequent reason for calling for help (8% of calls). The most seriously ill patients require the dispatch of specialized teams capable of initiating respiratory support in order to reduce the morbidity and mortality of these patients. In France, these teams are medicalized by an emergency physician within the Mobile Emergency Resuscitation Services (SMUR). This is only rarely the case outside France, where specialized paramedical teams ("advanced life support paramedic teams") can be dispatched. Apart from their role of initiating possible respiratory support, these teams (SMUR or paramedics) can initiate a diagnostic approach and therapeutics related to the suspected origin of dyspnea. However, there are many diagnoses that can cause dyspnea, and the diagnostic process can be complex. The most common diagnoses described in the prehospital population are: bacterial pneumonia, acute heart failure, and exacerbation of COPD or asthma or pulmonary embolism. Each of these diagnoses requires specific drug treatment, guided by international recommendations. Inappropriate treatment of these pathologies (overtreatment or undertreatment) is common and associated with excess intrahospital mortality.

Pleuropulmonary ultrasound (PUS) has shown very interesting diagnostic performance in the intrahospital setting for diagnoses of interest in dyspnea. This performance also appears good in the prehospital setting. In the intrahospital setting, PUS appears to improve the diagnostic approach and appropriate treatments for dyspnea. In the prehospital setting, however, data on this subject are scarce or of limited quality according to the most recent meta-analysis, while the use of this technique is becoming increasingly common in standardized patient care. In addition, the most recent work on the subject included patients in a non-medicalized prehospital system. The use of PUS would allow paramedics to increase the rate of appropriate treatment from 14% to 53%. However, the rate of appropriate treatment expected by a medicalized team is expected to be 62%, and the diagnostic performance of physicians in PUS is probably higher than that of paramedics. These data must therefore be consolidated in a French system before being the subject of higher-level recommendations. The systematic use of PUS during prehospital engagement of a SMUR for dyspnea also may improves the rate of appropriate treatment, even in a context of medicalization of the initial care of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Treated by a prehospital emergency medical service
* For dyspnea with signs of severity, the following are the following:

  * SpO2 < 90% in AA or O2 required to maintain SpO2 ≥ 90% and
  * RR > 25 cycles/min

Exclusion Criteria:

* Opposition to inclusion
* Need for immediate intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the emergency room for dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of pre-hospital EPP on the rate of appropriate treatments offered. | from the inclusion of the patient until the time he or she leaves the hospital, assessed up 52 weeks, whichever came first
  Therapeutic adequacy at the final diagnosis before and after completion of the PUS.
  Therapeutic adequacy and inadequacy are defined based on the treatment proposed before and after completion of the PUS, compared to the final diagnosis at hospital discharge. The following are considered inadequate:
  * In a patient on a pulmonary embolism (PE):
  * Prescribing beta-agonists or antibiotics (unless septic)
  * Not prescribing diuretics and nitrates if SBP > 140 mmHg
  * In a patient with decompensated COPD:
  * Prescribing diuretics
  * Not prescribing beta-agonists
  * In a patient with a pulmonary infection:
  * Prescribing diuretics
  * Not prescribing antibiotics
  * In a patient with a pulmonary embolism:
  * Not prescribing curative doses of anticoagulation In the case of multiple diagnoses (e.g., transfer to a PE due to pneumonia), only treatments that are inadequate for each diagnosis will be considered inadequate.

SECONDARY OUTCOMES:
Evaluation of the impact of PUS carried out in prehospital settings on the diagnostic process. | from the inclusion of the patient until the time he or she leaves the hospital, assessed up 52 weeks, whichever came first
  correct diagnosis(es) before and after PUS compared to the final diagnosis upon discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Marchetto, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Pôle Médecine d'Urgence Hôpital Purpan Pavillon Louis Lareng Place Docteur Baylac, Toulouse, France

IPD SHARING:
Plan to Share IPD: No